INFORMED CONSENT FOR PARTICIPATION IN THE CERTIFIED CLINICAL STUDY:

"Relevance of endometrial compaction in secretory phase in natural cycle for euploid embryo transfer"

## 1. INFORMATIVE DOCUMENT

We would like to propose you participate voluntarily in the clinical study entitled "Relevance of endometrial compaction in secretory phase in natural cycle for euploid embryo transfer"

With this study, we intend to deepen our understanding of the endometrial changes after ovulation in patients undergoing embryo transfer in natural cycle, investigating whether there is an association between changes in post-ovulatory endometrial thickness and pregnancy rate.

It is a non-intervention study; therefore, it does <u>NOT imply any change in your medical treatment nor</u> <u>does it entail any risk for you,</u> aspects of it will simply be analysed, and as the only additional intervention, a transvaginal ultrasound would be performed to assess the endometrium before the transfer.

If the treatment results in pregnancy, after delivery we may contact you by phone to inform us about the evolution of the pregnancy.

Your contribution is completely anonymous, confidential, and voluntary. It can be revoked at any time. This study complies with Organic Law 3/2018 of December 5<sup>th</sup> on the protection of personal data and guaranteed of digital rights, with the ethical conditions, having been approved for completion after evaluation by the Research Ethics Committee of Hospital de San Juan of Alicante.

The promoter and sole funder of this study is the Instituto Bernabeu, and it will be carried out exclusively in our centres, the main researcher being Dra. Esperanza de la Torre.

If you have any questions or comments related to the conduct of research, you can contact the investigators:

Dra. Esperanza de la Torre Pérez Ginecóloga especialista en Reproducción Asistida. Instituto Bernabeu Madrid (+34 918 333 882)

## 2. CONSENT DOCUMENT

| Me, | with passport number | <br>of legal | age, | consent | to: |
|---|---|---|---|---|---|
| participate in the research called: | | | | | |

"Relevance of endometrial compaction in secretory phase in natural cycle for euploid embryo transfer"

I have read the document, which includes clear and precise information from the investigation, regarding:

- o Main objective of the study
- o Mode of participation
- o Voluntariness
- Risks and benefits
- o Have a right to know the results
- O Have a right to withdraw from the study at any time, without having to give explanations or having an impact on my medical care
- Confidentiality
- o Information from the researcher, the Promoter, and the Scientific Ethics Committee

I have understood the statements enclosed in the document and the need to record my consent, for which I sign it freely and voluntarily, receiving on the spot a copy of this document already signed.

I talked to the Medical Team, who provided me all the information and I have been able to ask questions.

I agree to provide data on how my pregnancy has progressed and my baby's health after delivery.